CLINICAL TRIAL: NCT00665977
Title: Effect of Heated Humidity With Thermosmart™ Compared to an Intranasal Steroid in Improving Compliance and Nasal Symptoms in Patients Using Continuous Positive Airway Pressure
Acronym: Thermosmart
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clayton Sleep Insititute (Industry)
Responsible Party: Eric Powell, PhD, Clayton Sleep Institute, LLC
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F & P 07-004
Record Dates: First submitted 2008-02-07; First posted 2008-04-24 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Obstructive Sleep Apnea; Nasal Congestion; Sinus Congestion
Keywords: Obstructive Sleep Apnea; Nasal Congestion; Sinus congestion
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nasal Obstruction | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Sham Comparator): To enter into the single-blind placebo phase, subjects will be setup with a Fisher & Paykel 604 CPAP unit with a heated humidifier and "deactivated" Thermosmart™ tube, thus, only traditional heated humidity will be available. The deactivated unit will still "appear" to function with intact heated humidity settings. The CPAP machine will be set to the patient's prescribed pressure. Subjects will also be given a nasal steroid spray placebo and instructed to deliver one spray in each nostril daily.
  Interventions: Device: Placebo Arm
- Double Blind Treatment Group 2 (Active Comparator): Visit 3 will be identical to visit 2, with the exception being the crossover of double-blind treatment. Subjects will now receive the Fisher & Paykel 604 CPAP machine with traditional heated humidity and a deactivated Thermosmart™ tube set to their prescribed pressure. Subjects will also be given the nasal steroid Nasacort AQ (triamcinolone acetonide) at a dosage of 220 mcg. They will be instructed to deliver two sprays in each nostril daily. Once again, phone follow-up will be made 7-10 days after the visit to assess compliance with study procedures and adverse events.
  Interventions: Drug: Placebo Device & Nasacort
- Double Blind Treatment Goup 1 (Active Comparator): a Fisher & Paykel 604 CPAP machine with Thermosmart™ heated humidity set at their prescribed pressure. Subjects will also be given nasal steroid placebo (purified water) and instructed to deliver two sprays in each nostril daily
  Interventions: Drug: Thermosmart & placebo

INTERVENTIONS:
Drug: Thermosmart & placebo — a Fisher & Paykel 604 CPAP machine with Thermosmart™ heated humidity set at their prescribed pressure. Subjects will also be given nasal steroid placebo (purified water) and instructed to deliver two sprays in each nostril daily
  Arms: Double Blind Treatment Goup 1
Drug: Placebo Device & Nasacort — Visit 3 will be identical to visit 2, with the exception being the crossover of double-blind treatment. Subjects will now receive the Fisher & Paykel 604 CPAP machine with traditional heated humidity and a deactivated Thermosmart™ tube set to their prescribed pressure. Subjects will also be given the nasal steroid Nasacort AQ (triamcinolone acetonide) at a dosage of 220 mcg. They will be instructed to deliver two sprays in each nostril daily. Once again, phone follow-up will be made 7-10 days after the visit to assess compliance with study procedures and adverse events.
  Arms: Double Blind Treatment Group 2
Device: Placebo Arm — To enter into the single-blind placebo phase, subjects will be setup with a Fisher & Paykel 604 CPAP unit with a heated humidifier and "deactivated" Thermosmart™ tube, thus, only traditional heated humidity will be available. The deactivated unit will still "appear" to function with intact heated humidity settings. The CPAP machine will be set to the patient's prescribed pressure. Subjects will also be given a nasal steroid spray placebo and instructed to deliver one spray in each nostril daily.
  Arms: A

SUMMARY:
1. CPAP compliance will be significantly higher in both the heated humidity with Thermosmart™ and the nasal steroid phases compared to the double placebo phase.
2. CPAP compliance will be comparably improved in the heated humidity with Thermosmart™ phase versus the nasal steroid phase.
3. Improvement in nasal symptoms in using CPAP will be significantly improved in both the heated humidity with Thermosmart™ and the nasal steroid phases compared to the double placebo phase, and comparable between the heated humidity with Thermosmart™ phase versus the nasal steroid phase.
4. Secondary to improvements in CPAP compliance, measures of daytime functioning and quality of life will improve in the heated humidity with Thermosmart™ versus double placebo.

DETAILED DESCRIPTION:
Eligible participants will undergo this double-blind, placebo controlled, single-blind double placebo run-in, crossover trial to determine the efficacy of heated humidity with Thermosmart™ in improving compliance and nasal symptoms in patients using CPAP versus a nasal steroid and placebo (heated humidity, nasal steroid placebo) phases. After successful screening, participants will undergo a two week single-blind double placebo run-in phase using heated humidity and a nasal steroid placebo. The double-blind treatment phase will last a total of six weeks. Participants will undergo both phases: three weeks using heated humidity with Thermosmart™ and nasal steroid placebo and three weeks using a nasal steroid with a heated humidifier. Treatment phases will be counterbalanced. Study participation will last a total of 8 weeks from screening to completion of double-blind treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Diagnosis of obstructive sleep apnea (OSA) with apnea/hypopnea index (AHI) > 15/hr
* Currently using CPAP therapy and within 3 weeks to 12 months of initial CPAP titration
* Based on the CPAP nasal symptom questionnaire, a score of at least 3 (sometimes) for at least one of the following nasal symptoms related to their sleep apnea and CPAP usage: nasal congestion, runny nose, sneezing, or nasal irritation
* Willingness to tolerate and continue therapy with nCPAP
* Successfully titrated on nCPAP in a sleep center to a pressure between 6-16 cmH2O
* Willingness to comply and complete study related procedures
* Fluent in the English language

Exclusion Criteria:

* Co-morbid medical condition that is either medically significant and unstable, would interfere with the patient's ability to routinely use CPAP, or is a contraindication for use of a nasal steroid
* Women who are pregnant or who may potentially become pregnant during the course of the research trial.
* CPAP compliance over the past three weeks at screening > 5 hours/night, suggesting no compromised CPAP usage due to adverse nasal symptoms
* Wake resting SaO2 < 90%
* Currently using Bi-Level therapy, supplemental oxygen with CPAP therapy, or using a pressure outside inclusion criteria
* Currently using a Full-Face mask for CPAP therapy
* Current or prior use of the Fisher Paykel 604 CPAP machine with Thermosmart™ heated humidity.
* Patients who were never prescribed a heated humidifier with their CPAP machine (i.e. no humidifier or passover humidifier).
* Intranasal steroid treatment within the previous six months. Patient's currently taking intranasal steroid treatment cannot wash-out of steroid treatment to be included nor if patients have used nasal steroid treatment while on CPAP therapy
* Current upper airway tract infection, influenza, respiratory infection at time of screening or nasal surgery within 90 days of screening
* Prior surgical intervention for obstructive sleep apnea
* Currently taking medications that would be contraindicated to using a nasal steroid. Patients taking hypnotic or wake promoting therapy can participate if they have been on a stable dose prior to CPAP therapy and willing to maintain current dose as prescribed.
* Shift or rotating shift workers or individuals who routinely cannot contribute at least 6 hours/night to sleep/attempting therapy
* Additional sleep disorder that would interfere with routine use of CPAP

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Although an exact & universal definition of CPAP compliance has not been determined. Compliance will be tracked by the CPAP unit and downloaded into an analysis program for review at each visit. | 8 weeks

SECONDARY OUTCOMES:
Nasal Symptom Assessment, Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire, PSQI, Clayton Daytime Fatigue Scale, ESS, FSS, FOSQ, Actigraphy, Sleep, and Diary/Daily Assessments | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Powell, PhD, Principal Investigator — St. Louis University
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States